CLINICAL TRIAL: NCT04240002
Title: A Phase 1/2, Multicenter, Open-Label, Single Arm, Dose Escalation and Expansion Study of Gilteritinib (ASP2215) Combined With Chemotherapy in Children, Adolescents and Young Adults With FMS-like Tyrosine Kinase 3 (FLT3)/Internal Tandem Duplication (ITD) Positive Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: A Study of Gilteritinib (ASP2215) Combined With Chemotherapy in Children, Adolescents and Young Adults With FMS-like Tyrosine Kinase 3 (FLT3)/Internal Tandem Duplication (ITD) Positive Relapsed or Refractory Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to enrollment challenges.
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2215-CL-0603; 2018-002301-61 (EudraCT Number); 2024-512469-15 (Registry Identifier: EU CTIS)
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Results first posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia (AML); Acute Myeloid Leukemia With FMS-like Tyrosine Kinase 3 (FLT3) Mutation / Internal Tandem Duplication (ITD)
Keywords: ASP2215; Acute Myeloid Leukemia; FLT3; AML; gilteritinib
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — gilteritinib; fludarabine; Cytarabine; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Gilteritinib 2 mg/kg/day (Escalation Phase) (Experimental): Participants aged 2 years to less than 21 years with relapsed/refractory (R/R) FLT3 ITD and/or TKD Acute Myeloid Leukemia (AML) received 2 cycles (Cycle [C] 1 and C2) induction therapy with gilteritinib in combination with FLAG [fludarabine, cytarabine and granulocyte colony-stimulating factor (G-CSF)] chemotherapy. Gilteritinib tablet was administered at a starting dose of 2 milligrams/kilogram/day (mg/kg/day) (maximum 120 mg/day) orally once daily (QD) from days 8 to 21. FLAG regimen consisted of fludarabine: 30 milligrams per square meter (mg/m^2) per day intravenously (IV) from day 1 to day 5; cytarabine: 2000 mg/m^2 per day IV from day 1 to day 5; G-CSF (filgrastim): 5 micrograms per kilogram (μg/kg) per day subcutaneously (SC) or IV from day -1 to day 5. Each cycle = 28 days.
  Interventions: Drug: gilteritinib; Drug: fludarabine; Drug: cytarabine; Drug: granulocyte colony-stimulating factor (G-CSF)

INTERVENTIONS:
Drug: gilteritinib — Administered orally.
  Other Names: ASP2215
Drug: fludarabine — Administered by intravenous (IV) infusion
Drug: cytarabine — Administered by intravenous (IV) infusion
Drug: granulocyte colony-stimulating factor (G-CSF) — Administered by subcutaneous injection

SUMMARY:
The purpose of the phase 1 portion (dose escalation) of the study was to establish an optimally safe and biologically active recommended phase 2 dose (RP2D) and/or to determine maximum tolerated dose (MTD) for gilteritinib in sequential combination with fludarabine, cytarabine and granulocyte colony-stimulating factor (FLAG). The purpose of the phase 2 portion (dose expansion) was to determine complete remission (CR) rates and composite complete remission (CRc) rates after two cycles of therapy. The study also assessed safety, tolerability and toxicities of gilteritinib in combination with FLAG, evaluated FLT3 inhibition, assessed pharmacokinetics (PK), performed serial measurements of minimal residual disease, obtained preliminary estimates of 1-year event free survival (EFS) and overall survival (OS) rate and assessed the acceptability as well as palatability of the formulation.

One cycle was defined as 28 days of treatment. A participant completing 1 or 2 treatment cycles in phase 1 or 2 had the option to participate in long term treatment (LTT) with gilteritinib (for up to 2 years).

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged ≥ 6 months and < 21 years of age* at the time of signing informed consent and/or assent, as applicable.

  * *For phase 2: Enrollment of subjects from 6 months to less than 1 year and 1 year to less than 2 years will be dependent on the establishment of recommended phase 2 dose (RP2D) in the respective age groups during phase 1.
* Subject has a diagnosis of acute myeloid leukemia (AML) according to The French-American-British (FAB) classification with ≥ 5% blasts in the bone marrow, with or without extramedullary disease (except subjects with active central nervous system [CNS] leukemia).

  * In the phase 1 portion of the study, subject must be in first or greater relapse or refractory to induction therapy with no more than 1 attempt at remission induction (up to 2 induction cycles).
  * For the phase 2 portion of the study, subject must be in refractory to or at the first hematologic relapse after first-line remission induction AML therapy (up to 2 induction cycles).
* Subject has fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

  * Myelosuppressive chemotherapy:

    * For subject who relapses while receiving cytotoxic therapy, at least 21 days must have elapsed since the completion of cytotoxic therapy and prior to screening, unless the subject has recovered earlier than 21 days.
    * Cytoreduction with the following can be initiated and continued for up to 24 hours prior to the start of systemic protocol therapy (cycle 1 day -1).

      * hydroxyurea,
      * low dose cytarabine (100 mg/m^2 per dose once daily for 5 days) or
      * other low dose/maintenance therapies as per local site practice.
    * Subject who has received other FLT3 inhibitors (e.g., lestaurtinib, sorafenib, etc) is eligible for this study.
  * Hematopoietic growth factors: at least 7 days must have elapsed since the completion of therapy with a growth factor and prior to screening.
  * Biologic (anti-neoplastic agent): at least 7 days must have elapsed since the completion of therapy with a biologic agent and prior to screening. For agents that have known adverse events (AEs) occurring beyond 7 days after administration, this period must be extended beyond the time during which AEs are known to occur.
  * X-ray treatment (XRT):

    * 14 days must have elapsed for local palliative XRT for CNS chloromas and prior to screening; no washout period is necessary for other chloromas;
    * Prior to screening, 90 days must have elapsed if the subject had a prior traumatic brain injury or has received craniospinal XRT.
* For subject undergoing hematopoietic stem cell transplant (HSCT), at least 90 days must have elapsed since HSCT and subject must not have active graft-versus-host disease (GVHD).
* Subject has Karnofsky score ≥ 50 (if the subject is of ≥ 16 years of age) or Lansky score of ≥ 50 (if the subject is < 16 years of age). A score < 50 is acceptable if related to the subject's leukemia.
* Subject must meet the following criteria as indicated on the clinical laboratory tests.

  * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x upper limit normal (ULN) for age
  * Total serum bilirubin ≤ 1.5 x ULN for age
  * Estimated glomerular filtration rate of > 60 mL/min/1.73 m^2.
* A female subject is eligible to participate if she is not pregnant and at least 1 of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * WOCBP who agrees to follow the contraceptive guidance throughout the treatment period and for at least 180 days after the final study drug administration.
* Female subject must agree not to breastfeed starting at Screening, and throughout the study period and for 60 days after the final study drug administration.
* Female subject must not donate ova starting at Screening and throughout the study, and for 180 days after the final study drug administration.
* A male subject with female partner(s) of childbearing potential must agree to use contraception during the treatment period and for at least 180 days after the final study drug administration.
* A male subject must not donate sperm during the treatment period and for at least 120 days after the final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study period and for 180 days after the final study drug administration.
* Subject and subject's parent(s) or legal guardian agrees not to participate in another interventional study while on treatment.
* Live Vaccines - At least 6 weeks must have elapsed since the administration of the last dose of a live vaccine and prior to the initiation of study treatment (cycle 1, day -1)
* Phase 1: Subject is positive for FLT3 (ITD and/or tyrosine kinase domain [TKD]) mutation in bone marrow or blood as determined by the local institution.
* Phase 2: Subject is positive for the FLT3 (ITD) mutation in bone marrow or blood as determined by the local institution.

Exclusion Criteria:

* Subject has active CNS leukemia.
* Subject has uncontrolled or significant cardiovascular disease, including:

  * Diagnosed or suspected congenital long QT syndrome or any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de Pointes (TdP)); any history of arrhythmia will be discussed with the sponsor prior to subject's entry into the study
  * Prolonged Fridericia's Correction Formula (QTcF) interval on pre-entry electrocardiogram (ECG) (≥ 450 ms)
  * Any history of second or third degree heart block (may be eligible if the subject currently has a pacemaker)
  * Heart rate < 50 beats/minute on pre-entry ECG
  * Uncontrolled hypertension
  * Complete left bundle branch block
* Subject has systemic fungal, bacterial, viral or other infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment. The subject needs to be off pressors and have negative blood cultures for 48 hours.
* Subject is receiving or plans to receive concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
* Subject has active clinically significant GVHD or is on treatment with immunosuppressive drugs for treatment of active GVHD, with the exception of subjects being weaned from systemic corticosteroids where the subject is receiving ≤ 0.5 mg/kg of prednisone (or equivalent) daily dose for prior GVHD. Subject has received calcineurin inhibitors within 4 weeks prior to screening, unless used as GVHD prophylaxis.
* Subject has active malignant tumors other than AML.
* Subject has any significant concurrent disease, illness, psychiatric disorder or social issue that would compromise subject safety or compliance; interfere with consent, study participation, follow-up or interpretation of study results.
* Subject has hypokalemia and/or hypomagnesemia at Screening (defined as values below institutional lower limit of normal [LLN]). Repletion of potassium and magnesium levels during the screening period is allowed.
* Subject requires treatment with concomitant drugs that are strong inducers of cytochrome P450 (CYP)3A/P-glycoprotein (P-gp).
* Subject is known to have human immunodeficiency virus infection.
* Subject has active hepatitis B or C, or other active hepatic disorder.

  * Subjects with positive hepatitis B surface antigen (HBsAg) or detectable hepatitis B DNA are not eligible.
  * Subjects with negative HBsAg, positive hepatitis B core antibody and negative hepatitis B surface antibody will be eligible if hepatitis B DNA is undetectable.
  * Subjects with antibodies to hepatitis C virus will be eligible if hepatitis C RNA is undetectable.
* Subject must wait for at least 5 half-lives after stopping therapy with any investigational agent and before starting gilteritinib.
* Subject has a known or suspected hypersensitivity to gilteritinib, cytarabine, fludarabine, granulocyte colony-stimulating factor (G-CSF) or any components of the formulation used.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (7):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States
- Site DE49004, Essen, North Rhine-Westphalia, Germany
- SIte IT39001, Roma, Italy
- Site ES34001, Barcelona, Spain
- United Kingdom (3):
  - Site GB44001, Birmingham
  - Site GB44005, Cardiff
  - Site UK44007, Sutton

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Abematsu T, Nishikawa T, Shiba N, Iijima-Yamashita Y, Inaba Y, Takahashi Y, Nakagawa S, Kodama Y, Okamoto Y, Kawano Y. Pediatric acute myeloid leukemia co-expressing FLT3/ITD and NUP98/NSD1 treated with gilteritinib plus allogenic peripheral blood stem cell transplantation: A case report. Pediatr Blood Cancer. 2021 Nov;68(11):e29216. doi: 10.1002/pbc.29216. Epub 2021 Jul 10. No abstract available. PMID 34245496
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/2215-CL-0603
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14562&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants positive for FMS-like tyrosine kinase 3 (FLT3) [internal tandem duplication (ITD) and/or tyrosine kinase domain (TKD)] mutation in bone marrow or blood and positive for the FLT3 (ITD) mutation in bone marrow or blood were enrolled for phase 1 and phase 2 respectively.
Pre-assignment Details: The sponsor decided not to open the phase 2 extension part of the study and terminated the study after completion of the phase 1 dose escalation part for Group 1, hence, no participants were enrolled for dose escalation groups 2 and 3. The decision to terminate the study was based upon enrollment challenges due to the rarity of Relapsed or Refractory Acute Myeloid Leukemia (R/R AML) in children and not related to any safety or efficacy issues.
Period: Overall Study
Arm/Group | Gilteritinib 2 mg/kg/Day (Escalation Phase)
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all enrolled participants who received at least one dose of treatment regimen.
Groups:
- Gilteritinib 2 mg/kg/Day (Escalation Phase): Participants aged 2 years to less than 21 years with R/R FLT3 ITD and/or TKD AML received 2 cycles (C1 and C2) induction therapy with gilteritinib in combination with FLAG (fludarabine, cytarabine and G-CSF) chemotherapy. Gilteritinib tablet was administered at a starting dose of 2 mg/kg/day (maximum 120 mg/day) orally QD from days 8 to 21. FLAG regimen consisted of fludarabine: 30 mg/m^2 per day IV from day 1 to day 5; cytarabine: 2000 mg/m^2 per day IV from day 1 to day 5; G-CSF (filgrastim): 5 μg/kg per day SC or IV from day -1 to day 5. Each cycle = 28 days.
Arm/Group | Gilteritinib 2 mg/kg/Day (Escalation Phase)
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.9 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Percent Inhibition of Phosphorylated FMS-like Tyrosine Kinase 3 (FLT3) [Mean (Standard Deviation); unit: Percentage of pFLT3] — Baseline values were normalized such that each participant's baseline measurement of phosphorylated FLT3 (pFLT3) was set to 100%. All subsequent timepoint measurements were expressed as a percentage relative to this normalized baseline. Actual observed baseline values were not available. No additional statistical adjustments were applied beyond normalization
  Percentage of pFLT3 | 100.00 (0.00)

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD) of Gilteritinib
Description: MTD reflects the highest dose that did not cause a Dose Limiting Toxicity (DLT).DLT:any Grade ≥3 non-hematologic/extramedullary toxicity with the following exceptions that occurred during the DLT observations like alopecia, anorexia, or fatigue, grade 3 vomiting or diarrhea that resolved(with or without supportive care) to ≤ grade 2 within 48 hours, grade 3 nausea that resolved(with or without supportive care) to ≤ grade 2 within 7 days, grade 3 elevation in total bilirubin (TBL) that is asymptomatic and that returned to ≤ grade 2 elevation within 7 days, grade 3 elevation in hepatic transaminases[alanine aminotransferase (ALT/SGPT) aspartate aminotransferase (AST/SGOT) and gammaglutamyl transferase (GGT)] or Alkaline Phosphatase (ALP) level that returns to ≤ grade 2 elevation within 14 days, grade 3 fever with neutropenia, with/without infection, grade 3 infection/grade 4 infections expected as direct complication of cytopenia due to active underlying leukemia, grade 3 mucositis.
Time Frame: C1D1 up to day 28
Population: FAS
Measure: Number; unit: mg/kg/day
Arm/Group | Gilteritinib 2 mg/kg/Day (Escalation Phase)
Number analyzed (Participants) | 9
mg/kg/day | 2

2. Primary Outcome: Phase 1: Recommended Phase 2 Dose (RP2D) of Gilteritinib
Description: The RP2D was a safe dose of gilteritinib that demonstrated sufficient activity.
Time Frame: C1D1 up to day 28
Population: FAS
Measure: Number; unit: mg/kg/day
Arm/Group | Gilteritinib 2 mg/kg/Day (Escalation Phase)
Number analyzed (Participants) | 9
mg/kg/day | 2

3. Primary Outcome: Phase 2: Complete Remission (CR) Rate
Description: CR rate was defined as the number of participants with best response of CR divided by the number of participants in the analysis population. CR was defined as a morphologically leukemia-free state post-baseline and had absolute neutrophil count (ANC) >= 1 x 10^9/L, platelet count >= 100 x 10^9/L and normal marrow differential with < 5% blasts. and were red blood cell (RBC) and platelet transfusion independent (defined as 1 week without RBC transfusion and 1 week without platelet transfusion). There should be no evidence of extramedullary leukemia and no evidence of Auer rods. The blast counts in peripheral blood must be <= 2%. Derived and investigator-assessed responses are reported.
Time Frame: From date of randomization to end of induction (induction= 1-2 cycles, each cycle = 28 days)
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Gilteritinib 2 mg/kg/Day (Escalation Phase)
Number analyzed (Participants) | 9
Percentage of Participants
  Derived | 33.3 [7.5 to 70.1]
  Investigator | 33.3 [7.5 to 70.1]

4. Primary Outcome: Phase 2: Composite CR (CRc) Rate
Description: CRc was defined as participants who achieved either CR, complete remission with incomplete platelet recovery (CRp) or complete remission with incomplete hematologic recovery (CRi) at the visit. CR was defined as a morphologically leukemia-free state post-baseline and had ANC >= 1 x 10^9/L, platelet count >= 100 x 10^9/L and normal marrow differential with < 5% blasts. and were RBC and platelet transfusion independent (defined as 1 week without RBC transfusion and 1 week without platelet transfusion). There should be no evidence of extramedullary leukemia and no evidence of Auer rods. The blast counts in peripheral blood must be <= 2%. CRp was defined as met all CR criteria except incomplete platelet recovery (< 100x10^9/L). CRi was defined as met all CR criteria, except for incomplete hematological recovery with residual neutropenia < 1x10^9/L with or without complete platelet recovery. Derived and investigator-assessed responses are reported.
Time Frame: From date of randomization to end of induction (induction= 1-2 cycles, each cycle = 28 days)
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Gilteritinib 2 mg/kg/Day (Escalation Phase)
Number analyzed (Participants) | 9
Percentage of Participants
  Derived | 66.7 [29.9 to 92.5]
  Investigator | 55.6 [21.2 to 86.3]

5. Primary Outcome: Duration of CR
Description: Duration of CR was defined as the time from the date of first CR until the date of documented relapse for participants who achieved CR. CR was defined as a morphologically leukemia-free state post-baseline and had ANC >= 1 x 10^9/L, platelet count >= 100 x 10^9/L and normal marrow differential with < 5% blasts, and were RBC and platelet transfusion independent (defined as 1 week without RBC transfusion and 1 week without platelet transfusion). There should be no evidence of extramedullary leukemia and no evidence of Auer rods. The blast counts in peripheral blood must be <= 2%. Relapse was defined as a reappearance of leukemic blasts in the peripheral blood or >= 5% blasts in the bone marrow aspirate (BMA) not attributable to any other cause or reappearance or new appearance of extramedullary leukemia. Duration of CR was estimated using the Kaplan-Meier method.
Time Frame: From the date of first CR until the date of documented relapse for participants who achieved CR (Maximum duration: 28 months)
Population: FAS population included participants who achieved CR.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Gilteritinib 2 mg/kg/Day (Escalation Phase)
Number analyzed (Participants) | 3
days | NA [55.00 to NA] — Median and upper limit of the confidence interval was not estimable, due to insufficient number participants with events.

6. Primary Outcome: Phase 1: Number of Participants With Dose Limiting Toxicity (DLT) of Gilteritinib
Description: DLT: any Grade >=3 non-hematologic/extramedullary toxicity with the following exceptions that occurred during the DLT observation: Alopecia, anorexia, or fatigue. Grade 3 vomiting or diarrhea that resolved(with or without supportive care) to <= grade 2 within 48 hours. Grade 3 nausea that resolved(with or without supportive care) to <= grade 2 within 7 days. Grade 3 elevation in TBL that was asymptomatic and that returned to <= grade 2 elevation within 7 days. Grade 3 elevation in hepatic transaminases (ALT/SGPT, AST/SGOT) and GGT) or ALP level that returns to <= grade 2 elevation within 14 days. Grade 3 fever with neutropenia, with or without infection. Grade 3 infection or grade 4 infections expected as direct complication of cytopenia due to active underlying leukemia. Grade 3 mucositis.
Time Frame: C1D1 up to day 28
Population: Safety Analysis Set (SAF) included all enrolled participants who took at least 1 dose of treatment regimen. Participants who were DLT evaluable were analyzed.
Measure: Number; unit: Participants
Arm/Group | Gilteritinib 2 mg/kg/Day (Escalation Phase)
Number analyzed (Participants) | 8
Participants | 0

7. Secondary Outcome: Percent Change of Phosphorylated FMS-like Tyrosine Kinase 3 (FLT3)
Description: Plasma inhibitory assay (PIA) of phosphorylated FLT3 was conducted by comparing baseline and post-treatment samples. Inhibition was summarized at each time point. PIA assay assesses the target inhibition in plasma. Plasma was incubated with a cell line expressing the drug target, and inhibition was reported as percent change from baseline (normalized to 100%).
Time Frame: Baseline, predose on C1D15, C1D21, C2D8, C2D15, C2D21 and 4 to 6 hours post-dose on C1D21
Population: Pharmacodynamic Analysis Set (PDAS) included subset of the SAF for which sufficient pharmacodynamic measurements were collected. PDAS with available data was analyzed.
Measure: Mean (Standard Deviation); unit: Percent Change of pFLT3
Arm/Group | Gilteritinib 2 mg/kg/Day (Escalation Phase)
Number analyzed (Participants) | 9
Percent Change of pFLT3
  Cycle 1 Day 15 Pre-Dose | 15.00 (14.41)
  Cycle 1 Day 21 Pre-Dose: number analyzed (Participants) | 8
  Cycle 1 Day 21 Pre-Dose | 11.96 (11.85)
  Cycle 1 Day 21 4-6 Hours Post-Dose | 7.32 (9.14)
  Cycle 2 Day 8 Pre-Dose: number analyzed (Participants) | 3
  Cycle 2 Day 8 Pre-Dose | 63.97 (25.40)
  Cycle 2 Day 15 Pre-Dose: number analyzed (Participants) | 3
  Cycle 2 Day 15 Pre-Dose | 9.90 (2.95)
  Cycle 2 Day 21 Pre-Dose: number analyzed (Participants) | 3
  Cycle 2 Day 21 Pre-Dose | 6.03 (8.72)

8. Secondary Outcome: Gilteritinib Plasma Concentration
Description: Plasma samples were used for pharmacokinetic assessments.
Time Frame: Predose on C1D8, C1D15, C1D21, C2D15, and 4 to 6 hours post-dose on C1D21
Population: The pharmacokinetic analysis set (PKAS) included the administered population for which sufficient plasma concentration data was available to facilitate derivation of at least 1 pharmacokinetic parameter and for whom the time of dosing on the day of sampling was known. PKAS with available data was analyzed.
Measure: Mean (Standard Deviation); unit: nanogram (ng)/mL
Arm/Group | Gilteritinib 2 mg/kg/Day (Escalation Phase)
Number analyzed (Participants) | 9
nanogram (ng)/mL
  Cycle 1 Day 8 Pre-Dose: number analyzed (Participants) | 8
  Cycle 1 Day 8 Pre-Dose | 0 (0)
  Cycle 1 Day 15 Pre-Dose | 251.93 (202.55)
  Cycle 1 Day 21 Pre-Dose: number analyzed (Participants) | 8
  Cycle 1 Day 21 Pre-Dose | 225.25 (135.18)
  Cycle 1 Day 21 4-6 Hours Post-Dose | 439.00 (209.62)
  Cycle 2 Day 15 Pre-Dose: number analyzed (Participants) | 3
  Cycle 2 Day 15 Pre-Dose | 145.07 (67.09)

9. Secondary Outcome: Pharmacokinetics (PK) of Gilteritinib: Oral Clearance (CL/F)
Time Frame: Predose on C1D8, C1D15, C1D21, C2D15, and 4 and 6 hours post-dose on C1D21
Reporting Status: Not Posted, anticipated posting 2027-12

10. Secondary Outcome: PK of Gilteritinib: Apparent Volume of Distribution (Vd/F)
Time Frame: Predose on C1D8, C1D15, C1D21, C2D15, and 4 and 6 hours post-dose on C1D21
Reporting Status: Not Posted, anticipated posting 2027-12

11. Secondary Outcome: PK of Gilteritinib: Maximum Plasma Concentration (Cmax)
Time Frame: Predose on C1D8, C1D15, C1D21, C2D15, and 4 and 6 hours post-dose on C1D21
Reporting Status: Not Posted, anticipated posting 2027-12

12. Secondary Outcome: PK of Gilteritinib: Time to Observed Cmax (Tmax)
Time Frame: Predose on C1D8, C1D15, C1D21, C2D15, and 4 and 6 hours post-dose on C1D21
Reporting Status: Not Posted, anticipated posting 2027-12

13. Secondary Outcome: PK of Gilteritinib: Area Under the Concentration (AUC)
Time Frame: Predose on C1D8, C1D15, C1D21, C2D15, and 4 and 6 hours post-dose on C1D21
Reporting Status: Not Posted, anticipated posting 2027-12

14. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE could therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. TEAE was defined as an adverse event observed after starting administration of the study drug until 28 days from the last study treatment.
Time Frame: From first dose up to 28 days after last dose (maximum duration approximately 55 months)
Population: SAF
Measure: Number; unit: Participants
Arm/Group | Gilteritinib 2 mg/kg/Day (Escalation Phase)
Number analyzed (Participants) | 9
Participants | 9

15. Secondary Outcome: Event Free Survival (EFS)
Description: EFS was defined as the time from first study drug dose to documented relapse or death, whichever occurred first. If none of these events occurred, EFS was censored at the last relapse-free assessment. Relapse was defined as a reappearance of leukemic blasts in the peripheral blood or >= 5% blasts in the BMA not attributable to any other cause or reappearance or new appearance of extramedullary leukemia. EFS was estimated using the Kaplan-Meier method.
Time Frame: From first dose to documented relapse or death, whichever occurred first (maximum duration: 55 month)
Population: FAS
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Gilteritinib 2 mg/kg/Day (Escalation Phase)
Number analyzed (Participants) | 9
days | 123.00 [1.00 to NA] — Upper limit of the confidence interval was not estimable, due to insufficient number participants with events.

16. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of enrollment until the date of death from any cause (death date - enrollment date + 1). For a participant who was not known to have died by the end of study follow-up, OS was censored at the date of last contact (date of last contact - enrollment date + 1). OS was estimated using the Kaplan-Meier method.
Time Frame: From the date of enrollment until the date of death from any cause (maximum duration: 55 months)
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gilteritinib 2 mg/kg/Day (Escalation Phase)
Number analyzed (Participants) | 9
months | NA [4.80 to NA] — Median and upper limit of the confidence interval was not estimable, due to insufficient number participants with events.

17. Secondary Outcome: Number of Participants With Negative Minimal Residual Disease (MRD) Status
Description: MRD negative was defined as summed FLT3-ITD signal ratio of any post-baseline sample ≤10^(-4).
Time Frame: From baseline up to approximately 55 months
Population: The MRD Analysis Set (MAS) included a subset of the FAS for which participants enrolled, received at least 1 dose of the treatment regimen, and had at least 1 post-baseline sample with MRD data.
Measure: Number; unit: Participants
Arm/Group | Gilteritinib 2 mg/kg/Day (Escalation Phase)
Number analyzed (Participants) | 5
Participants | 4

18. Secondary Outcome: Percentage of Participants With MRD Negative Status in Relation to CR Rate
Description: MRD negative was defined as summed FLT3-ITD signal ratio of any post-baseline sample <=10^(-4). CR rate was defined as the number of participants with best response of CR divided by the number of participants in the analysis population. CR was defined as a morphologically leukemia-free state post-baseline and had ANC >= 1 x 10^9/L, platelet count >= 100 x 10^9/L and normal marrow differential with < 5% blasts. and were RBC and platelet transfusion independent (defined as 1 week without RBC transfusion and 1 week without platelet transfusion). There should be no evidence of extramedullary leukemia and no evidence of Auer rods. The blast counts in peripheral blood must be <= 2%. Derived and investigator-assessed responses are reported.
Time Frame: From baseline up to approximately 55 months
Population: MAS with available data was analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gilteritinib 2 mg/kg/Day (Escalation Phase)
Number analyzed (Participants) | 4
percentage of participants
  Derived | 75.0 [19.4 to 99.4]
  Investigator | 75.0 [19.4 to 99.4]

19. Secondary Outcome: Percentage of Participants With MRD Negative Status in Relation to CRc Rate
Description: MRD negative: summed FLT3-ITD signal ratio of any post-baseline sample <=10^(-4). CRc: participants who achieved either CR, complete remission with CRp or CRi at the visit. CR: morphologically leukemia-free state post-baseline and had ANC >= 1 x 10^9/L, platelet count >= 100 x 10^9/L and normal marrow differential with < 5% blasts. and were RBC and platelet transfusion independent. There should be no evidence of extramedullary leukemia and no evidence of Auer rods. The blast counts in peripheral blood must be <= 2%. CRp: all CR criteria except incomplete platelet recovery (< 100x10^9/L). CRi: met all CR criteria, except for incomplete hematological recovery with residual neutropenia < 1x10^9/L with or without complete platelet recovery. CRc rate: as number of participants with best response of CR divided by the number of participants in the analysis population. Derived and investigator-assessed responses are reported.
Time Frame: From baseline up to approximately 55 months
Population: MAS with available data was analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gilteritinib 2 mg/kg/Day (Escalation Phase)
Number analyzed (Participants) | 4
percentage of participants
  Derived | 100.0 [39.8 to 100.0]
  Investigator | 100.0 [39.8 to 100.0]

20. Secondary Outcome: Number of Participants With MRD Negative Status in Relation to OS
Description: MRD negative: summed FLT3-ITD signal ratio of any post-baseline sample ≤10^(-4). OS was defined as the time from the date of enrollment until the date of death from any cause (death date - enrollment date + 1). For a participant who was not known to have died by the end of study follow-up, OS was censored at the date of last contact (date of last contact - enrollment date + 1).
Time Frame: From baseline up to approximately 55 months
Population: MAS with available data was analyzed.
Measure: Number; unit: participants
Arm/Group | Gilteritinib 2 mg/kg/Day (Escalation Phase)
Number analyzed (Participants) | 4
participants | 1

21. Secondary Outcome: Number of Participants With Gilteritinib Acceptability and Palatability for Tablet
Description: Participants evaluated the taste of the study drug/tablets and indicated whether they would be willing (feeling) to take the study drug/tablets again by selecting one of the following categories: 'Like a lot,' 'Like a little,' 'Neither like nor dislike,' 'Dislike a little,' or 'Dislike a lot.'
Time Frame: C1D1, C1D8
Population: FAS with available data was analyzed.
Measure: Number; unit: Participants
Arm/Group | Gilteritinib 2 mg/kg/Day (Escalation Phase)
Number analyzed (Participants) | 7
Participants
  C1D8 Tastes: Like a lot: number analyzed (Participants) | 6
  C1D8 Tastes: Like a lot | 1
  C1D8 Tastes: Like a little: number analyzed (Participants) | 6
  C1D8 Tastes: Like a little | 2
  C1D8 Tastes: Neither like or dislike: number analyzed (Participants) | 6
  C1D8 Tastes: Neither like or dislike | 3
  C1D8 Tastes: Dislike a little: number analyzed (Participants) | 6
  C1D8 Tastes: Dislike a little | 0
  C1D8 Tastes: Dislike a lot: number analyzed (Participants) | 6
  C1D8 Tastes: Dislike a lot | 0
  C1D8 Feeling: Like a lot: number analyzed (Participants) | 6
  C1D8 Feeling: Like a lot | 3
  C1D8 Feeling: Like a little: number analyzed (Participants) | 6
  C1D8 Feeling: Like a little | 1
  C1D8 Feeling: Neither like or dislike: number analyzed (Participants) | 6
  C1D8 Feeling: Neither like or dislike | 2
  C1D8 Feeling: Dislike a little: number analyzed (Participants) | 6
  C1D8 Feeling: Dislike a little | 0
  C1D8 Feeling: Dislike a lot: number analyzed (Participants) | 6
  C1D8 Feeling: Dislike a lot | 0
  C1D21 Tastes: Like a lot | 1
  C1D21 Tastes: Like a little | 1
  C1D21 Tastes: Neither like or dislike | 5
  C1D21 Tastes: Dislike a little | 0
  C1D21 Tastes: Dislike a lot | 0
  C1D21 Feeling: Like a lot | 3
  C1D21 Feeling: Like a little | 1
  C1D21 Feeling: Neither like or dislike | 3
  C1D21 Feeling: Dislike a little | 0
  C1D21 Feeling: Dislike a lot | 0

ADVERSE EVENTS:
Time Frame: All Cause: From randomization up to end of study (maximum duration approximately 55 months) AE: From first dose up to 28 days after last dose (maximum duration approximately 55 months)
Description: SAF included all participants who took at least 1 dose of the treatment regimen.
Arm/Group | Gilteritinib 2 mg/kg/Day (Escalation Phase)
All-Cause Mortality (participants affected / at risk) | 4/9
Serious Adverse Events (participants affected / at risk) | 7/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilteritinib 2 mg/kg/Day (Escalation Phase) (N=9)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Pyrexia (General disorders) | 1 (2)
Graft versus host disease in eye (Immune system disorders) | 1 (1)
Graft versus host disease in liver (Immune system disorders) | 2 (2)
Graft versus host disease oral (Immune system disorders) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Device related bacteraemia (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Tooth abscess (Infections and infestations) | 1 (1)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilteritinib 2 mg/kg/Day (Escalation Phase) (N=9)
Anaemia (Blood and lymphatic system disorders) | 5 (41)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (9)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3)
Cardiac failure (Cardiac disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (5)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (7)
Nausea (Gastrointestinal disorders) | 5 (8)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (14)
Catheter site pain (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 6 (12)
Swelling face (General disorders) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Fungal foot infection (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (2)
Herpes zoster (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 1 (3)
Nasal herpes (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1)
Avulsion fracture (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (39)
Aspartate aminotransferase increased (Investigations) | 6 (20)
Blood bicarbonate decreased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 3 (6)
Blood creatinine increased (Investigations) | 2 (2)
Blood culture positive (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 3 (7)
Blood potassium decreased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (36)
Mean arterial pressure decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (4)
Oxygen saturation decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 3 (55)
White blood cell count decreased (Investigations) | 3 (11)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3)
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 (3)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (7)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (3)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (29)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (15)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (11)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (15)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (6)
Iron overload (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Hypotonia (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (2)
Presyncope (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Irritability (Psychiatric disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 4 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Axillary vein thrombosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated because of enrollment challenges due to the rarity of R/R AML in children and not related to any safety or efficacy issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT04240002/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT04240002/SAP_001.pdf